CLINICAL TRIAL: NCT01578629
Title: Human Blood Outcomes Following Tocotrienol Supplementation - NUTRITION Phase I and Phase IIA
Brief Title: NUTRITION: Natural Tocotrienol Against Ischemic Stroke Event
Acronym: NUTRITION
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andrew Slivka (Other)
Collaborators: Government of Malaysia (Unknown)
Responsible Party: Sponsor-Investigator, Andrew Slivka, MD, Professor of Neurology, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2011H0242
Record Dates: First submitted 2012-04-05; First posted 2012-04-17 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack (TIA)
Keywords: stroke; ischemia; TIA
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Stroke; Ischemia | interventions — Thrombin Time; Capsules; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Active Comparator): Healthy participants randomized into one of 6 groups that will take 4 capsules, twice a day of vitamin E tocotrienol (TCT) capsules ; Low Dose Aspirin or placebo capsule for 7 months.
  Interventions: Other: Vitamin E tocotrienol (TCT) capsules ; Low dose Aspirin; Other: Placebo vehicle control
- Hyperlipidemic (Active Comparator): hyperlipidemic patients randomized into one of 6 groups that will take 4 capsules, twice a day of Vitamin E Tocotrienol (TCT) capsules; Low Dose Aspirin or placebo vehicle control capsule for 7 months.
  Interventions: Other: Vitamin E tocotrienol (TCT) capsules ; Low dose Aspirin; Other: Placebo vehicle control

INTERVENTIONS:
Other: Vitamin E tocotrienol (TCT) capsules ; Low dose Aspirin — Vitamin E TCT capsules- 400-800 mg Aspirin- 81 mg
Other: Placebo vehicle control — vehicle control compared to Vitamin E TCT pills
  Other Names: placebo capsule

SUMMARY:
A natural form of vitamin E called tocotrienol (TCT), found in many common foods such as barley, decreases stroke size in animal models. Vitamin E has blood-thinning properties and lowers cholesterol, which make it a potential therapy for stroke prevention, though these effects are less well characterized for TCT. We plan to conduct two trials (I & IIA) to determine the effects of orally supplemented TCT on platelet function and cholesterol.

DETAILED DESCRIPTION:
A natural form of vitamin E called tocotrienol (TCT), found in many common foods such as barley, decreases stroke size in animal models. Vitamin E has blood-thinning properties and lowers cholesterol, which make it a potential therapy for stroke prevention, though these effects are less well characterized for TCT. We plan to conduct two trials (I & IIA) to determine the effects of orally supplemented TCT on platelet function and cholesterol. Phase I subjects will be healthy volunteers, recruited by an advertisement. Phase IIA subjects will be hyperlipidemic (having high cholesterol), and will be referred to us by their Wound Care Center Physicians. Patients will be randomized to receive placebo pills, (400 or 800 mg) TCT pills, low-dose 81 mg aspirin (commonly used for secondary prevention of stroke), or TCT and aspirin together. Potential subjects for Phase-I who meet study criteria and agree to participate will be in the study for 6 months and have the following study related procedures, blood draw total 4 times, tape stripping (non-invasive procedure), BMI, and blood pressure measurement at each visit (every month). Participants in Phase-IIA will have blood drawn a total of 6 times, tape stripping, BMI and blood pressure measurement and participants will be in the study for 13 months.

ELIGIBILITY:
Phase IA

Inclusion Criteria:

* Healthy subjects between 40 and 70 years of age
* No history of long-term vitamin E supplement (defined as daily oral tocopherol or tocotrienol supplementation greater than or equal to 6mos; within the past 5 years)
* No current vitamin E supplementation in multivitamin

Exclusion Criteria - (as self reported by potential participants during review of eligibility criteria with Research Nurse,)

* Evidence of heart disease as diagnosed by a physician by one or more of the following tests; EKG, chest x-ray, stress test, tilt table test, echocardiogram, coronary angiogram, electrophysiology test, CT heart scan, coronary MRI, pericardiocentesis
* High cholesterol (total cholesterol >240mg/dL, LDL>160mg/dL)
* Prior cancer diagnosis
* Pregnancy - To exclude the possibility of pregnant women entering the study or becoming pregnant during the study only post-menopausal women or women who have had hysterectomies or bilateral oophorectomies will be included.
* Breast feeding
* Smoker (Must have quit 5 or more years ago)
* Alcohol dependence (>4 drinks per day for more than 1yr anytime in the last 3 years)
* Medication exclusion criteria - current use or recent discontinuation (within last 28 days) of any medication including the following: anti-coagulants and blood-thinners (e.g., Warfarin), psychotropic medications including antipsychotics, mood-stabilizers (e.g., lithium, valproic acid, carbamazepine/tegretol); anti-depressants (tricyclics, SSRI's, MAOI's, nonselective MAOIs, Wellbutrin, St. John's Wort); anti-anxiety/anti-panic agents; anti-obsessive agents; prescription stimulants (e.g., Provigil, Ritalin); diet pills/anorectics; daily medication for chronic pain (e.g., opiates) or muscle spasms; daily use of over the counter stimulants in pill form (e.g., ephedrine); daily medication for asthma, Parkinson's disease medications (e.g., levodopa, methyldopa, apomorphine), smoking cessation medications (Wellbutrin/Zyban, Chantix/varenicline); statin use is not grounds for exclusion.

Phase IIA

Inclusion Criteria:

* Hyperlipidemic patients between 40 and 70 years of age currently taking statins
* LDL>130mg/dL
* TG>150mg/dL
* HDL<40mg/dL
* No history of long-term vitamin E supplement (defined as daily oral tocopherol or tocotrienol supplementation greater than or equal to 6mos; within the past 5 years)
* No current vitamin E supplementation in multivitamin

Exclusion Criteria:

* Evidence of heart disease as diagnosed by a physician by one or more of the following tests; EKG, chest x-ray, stress test, tilt table test, echocardiogram, coronary angiogram, electrophysiology test, CT heart scan, coronary MRI, pericardiocentesis
* Prior cancer diagnosis
* Currently taking blood thinners
* Pregnancy - To exclude the possibility of pregnant women entering the study or becoming pregnant during the study only post-menopausal women or women who have had hysterectomies or bilateral oophorectomy will be included.
* Breast feeding
* Smoking (Must have quit within the past 6 months)
* Alcohol dependence - (>4 drinks per day for more than 1yr anytime in the last 3 years)
* Medication exclusion criteria - current use or recent discontinuation (within last 28 days) of any medication including the following: anti-coagulants and blood-thinners (e.g., Warfarin), psychotropic medications including antipsychotics, mood-stabilizers (e.g., lithium, valproic acid, carbamazepine/tegretol); anti-depressants (tricyclics, SSRI's, MAOI's, nonselective MAOIs, Wellbutrin, St. John's Wort); anti-anxiety/anti-panic agents; anti-obsessive agents; prescription stimulants (e.g., Provigil, Ritalin); diet pills/anorectics; daily medication for chronic pain (e.g., opiates) or muscle spasms; daily use of over the counter stimulants in pill form (e.g., ephedrine); daily medication for asthma, Parkinson's disease medications (e.g., levodopa, methyldopa, apomorphine), smoking cessation medications (Wellbutrin/Zyban, Chantix/varenicline)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-03; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Platelet function panel | up to one year
  Blood draw followed by platelet aggregometry
Lipid profile | up to one year
  blood lipid panel including HDL, LDL, total cholesterol

SECONDARY OUTCOMES:
Tape Stripping Test | up to one year
  HPLC vitamin E analysis of tape strips for compliance

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio state University Medical Center, Columbus, Ohio, United States